CLINICAL TRIAL: NCT06400342
Title: Randomized Evaluation of Valve-In-Valve Versus Explantation for Failed TAVR (REVIVE-TAVR)
Brief Title: Randomized Evaluation for Failed TAVR
Acronym: REVIVE-TAVR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REVIVE-TAVR
Record Dates: First submitted 2024-03-25; First posted 2024-05-06 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Symptomatic Patients Who Have Had Transcatheter Heart Valve (THV) Failure; Prosthetic Valve Malfunction; Prosthesis Failure
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Subjects deemed eligible for both redo-TAVR and TAVR-explant by the Heart Team for the treatment of failed THV will be randomized on a 1:1 basis to either redo-TAVR or TAVR-explant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- TAVR-explant (Active Comparator): TAVR surgical explantation
  Interventions: Procedure: TAVR-explant
- Redo-TAVR (Active Comparator): TAV-in-TAV
  Interventions: Device: Redo-TAVR

INTERVENTIONS:
Procedure: TAVR-explant — Surgical explantation of failed THV followed by surgical aortic valve replacement and any other cardiac surgeries deemed necessary.
  Arms: TAVR-explant
Device: Redo-TAVR — Repeat transcatheter aortic valve implantation within a failed THV.
  Other Names: Valve-in-Valve, TAV-in-TAV
  Arms: Redo-TAVR

SUMMARY:
REVIVE TAVR is an acronym for the Randomized Evaluation of Valve-In-Valve versus Explantation for failed TAVR. This is a prospective, multicenter, global randomized trial investigating the safety and efficacy of reintervention for transcatheter heart valve (THV) failure by comparing redo-TAVR (TAV-in-TAV) with TAVR surgical explantation (TAVR-explant) in subjects who are suitable for both options in a real-world clinical setting

ELIGIBILITY:
Inclusion Criteria:

* Heart Team has confirmed eligibility for both TAVR-explant and redo-TAVR for failed THV
* Subject is symptomatic from their failed THV, as demonstrated by NYHA Functional Class ≥II
* Subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits
* Subject meets the legal minimum age to provide informed consent based on local regulatory requirements.

Exclusion Criteria:

* Ongoing sepsis, including active endocarditis;
* Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits);
* Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the subject from appropriate consent or adherence to the protocol required follow-up exams;
* Pregnancy or intent to become pregnant for the next 12 months;

Coronary obstruction risk:

- Patients at risk of coronary obstruction may be enrolled into the randomized cohort if the operators determine that redo-TAVR can be safely accomplished with leaflet modification or other coronary protection strategies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2034-05-01 (Estimated); Study Completion 2036-05-01 (Estimated)

PRIMARY OUTCOMES:
Composite: All-cause mortality, stroke, and rehospitalization for cardiovascular causes | 30 days
  Time to first event of any components of the composite endpoint.
Composite: All-cause mortality, stroke, and rehospitalization for cardiovascular causes | 12 months
  Time to first event of any components of the composite endpoint.

SECONDARY OUTCOMES:
All-cause mortality | 30 days
  Cardiovascular mortality, Valve-related mortality, Non-cardiovascular mortality
All-cause mortality | 12 months
  Cardiovascular mortality, Valve-related mortality, Non-cardiovascular mortality
Stroke | 30 days
Stroke | 12 months
Rehospitalization for cardiovascular causes | 30 days
Rehospitalization for cardiovascular causes | 12 months
Reintervention hospital length of stay (days) | 30 days
Cardiovascular mortality | 30 days
  Death meeting one of the following criteria:
  * related to heart failure, cardiogenic shock, bioprosthetic valve dysfunction, myocardial infarction, stroke, thromboembolism, bleeding, tamponade, vascular complication, arrhythmia or conduction system disturbances, cardiovascular infection (e.g. mediastinitis, endocarditis), or other clear cardiovascular cause
  * Intraprocedural death
  * Sudden death
  * Death of unknown cause
  Valve-related mortality
  - Death presumed to be related to bioprosthetic valve dysfunction
Cardiovascular mortality | 12 months
  Death meeting one of the following criteria:
  * related to heart failure, cardiogenic shock, bioprosthetic valve dysfunction, myocardial infarction, stroke, thromboembolism, bleeding, tamponade, vascular complication, arrhythmia or conduction system disturbances, cardiovascular infection (e.g. mediastinitis, endocarditis), or other clear cardiovascular cause
  * Intraprocedural death
  * Sudden death
  * Death of unknown cause
  Valve-related mortality
  - Death presumed to be related to bioprosthetic valve dysfunction
VARC-3 bleeding | 30 days
VARC-3 bleeding | 12 months
Vascular and access-related complications | 30 days
Vascular and access-related complications | 12 months
Cardiac structural complications | 30 days
Cardiac structural complications | 12 months
Other acute procedural and technical valve-related complications | 30 days
Other acute procedural and technical valve-related complications | 12 months
Conduction disturbance requiring permanent pacemaker implantation | 30 days
Conduction disturbance requiring permanent pacemaker implantation | 12 months
Acute kidney injury | 30 days
Acute kidney injury | 12 months
Myocardial infarction (adapted from 4th Universal, SCAI, and ARC-2 definitions) | 30 days
Myocardial infarction (adapted from 4th Universal, SCAI, and ARC-2 definitions) | 12 months
Bioprosthetic valve dysfunction (BVD) and failure (BVF) as defined by the Valve Academic Research Consortium (VARC)-3 Criteria. | 30 days
Bioprosthetic valve dysfunction (BVD) and failure (BVF) as defined by the Valve Academic Research Consortium (VARC)-3 Criteria. | 12 months
Echocardiographic assessment of prosthetic valve performance | 30 days
Echocardiographic assessment of prosthetic valve performance | 12 months
Change in NYHA class from Baseline | 30 days
Change in NYHA class from Baseline | 12 months
Change in Quality of life (KCCQ) from Baseline | 30 days
  The KCCQ has a 0-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Change in Quality of life (KCCQ) from Baseline | 12 months
  The KCCQ has a 0-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Technical Success | 30 days
  * Freedom from mortality
  * Successful access, delivery of the device and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Device Success (for Redo-TAVR) | 30 days
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve
Safety Composite Endpoints | 30 days
  * Early safety, which includes freedom from all-cause mortality, all stroke, VARC type 2-4 bleeding, major vascular, access-related or cardiac structural complication, acute kidney injury stage 3 or 4, moderate or severe aortic regurgitation, new permanent pacemaker due to procedure-related conduction abnormalities and surgery or intervention related to the device.
  * Clinical efficacy
  * Valve-related long-term clinical efficacy
Technical Success | 12 months
  Same as above (Technical Success outcome 34)
Device Success (for Redo-TAVR) | 12 months
  Same as above (Device Success (for Redo-TAVR) outcome 35)
Safety Composite Endpoints | 12 months
  Same as above (Safety Composite Endpoints outcome 36)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — MedStar Health Research Organization; Toby Rogers, MD, Study Chair — MedStar Health Research Organization; Thomas MacGillivray, MD, Study Chair — MedStar Health Research Organization; Michael Reardon, MD, Study Chair — MedStar Health Research Organization; Kalyan Chitturi, DO, Study Chair — MedStar Health Research Organization

IPD SHARING:
Plan to Share IPD: Undecided